CLINICAL TRIAL: NCT01436071
Title: A Randomised, Double-blind, Placebo-controlled (With Rescue Medication), Multi-centre Study to Evaluate the Efficacy and Safety of Inhaled Fluticasone Furoate in the Treatment of Persistent Asthma in Adults and Adolescents Not Currently Receiving Inhaled Corticosteroids
Brief Title: Clinical Study Evaluating Safety and Efficacy of Fluticasone Furoate in People With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115283
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone furoate 50mcg (Experimental): Inhalation powder delivered by Novel Dry Powder Inhaler
  Interventions: Drug: Fluticasone furoate 50mcg
- Placebo (Placebo Comparator): Inhalation powder delivered by Novel Dry Powder Inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone furoate 50mcg — Inhalation powder delivered by Novel Dry Powder Inhaler
  Arms: Fluticasone furoate 50mcg
Drug: Placebo — Inhalation powder delivered by Novel Dry Powder Inhaler
  Arms: Placebo

SUMMARY:
A randomised, double-blind, placebo-controlled (with rescue medication), multi-centre study to evaluate the efficacy and safety of inhaled fluticasone furoate in the treatment of persistent asthma in adults and adolescents not currently receiving inhaled corticosteroids

DETAILED DESCRIPTION:
This will be a multi-centre, randomised, placebo controlled (with rescue medication), double-blind, parallel group study. Subjects meeting all the inclusion criteria and none of the exclusion criteria during Visit 1 (Screening Visit) will enter a two week Run-in Period. Subjects failing screening will not be eligible for re-screening. During the run-in and double-blind treatment periods subjects will maintain an electronic daily diary to record morning and evening peak expiratory flow (PEF), asthma symptom score and rescue albuterol/salbutamol use. At Visit 2 (end of run-in/Randomisation Visit), subjects meeting the eligibility criteria will be randomised to either inhaled Fluticasone Furoate 50 mcg or inhaled placebo. In addition all subjects will be supplied with albuterol/salbutamol inhalation aerosol to use as required to treat symptoms. Subjects will attend 4 on-treatment visits at Visits 3, 4, 5, and 6 (Weeks 2, 4, 8 and 12 respectively). Subjects will receive treatment for 84 days (12 weeks). A follow-up contact will be performed 1-week after completing study medication (Visit 7). Subjects will participate in the study for up to a maximum of 15 weeks (including screening, treatment and follow-up contact).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Outpatient at least 12 years of age with diagnosis of asthma at least 12 weeks before first visit
* Both genders; females of child bearing potential must be willing to use appropriate contraception during the study
* Pre-bronchodilator FEV1 of at least 60% predicted
* FEV1 reversibility of at least 12% and 200mls
* Current asthma therapy that includes a non-corticosteroid controller and/or short-acting beta agonist

Exclusion Criteria:

* History of life-threatening asthma exacerbation within the past 10 years
* Asthma exacerbation requiring treatment with oral corticosteroids within the last 3 months or that required overnight hospital stay within 6 months
* Current or recent respiratory infection or current oral candida infection
* Presence of another significant respiratory disease or medical condition that is not controlled or that could affect subject safety or study outcome
* Known or suspected allergy to study drug or materials
* Taking another investigational medication or prohibited medication during the study
* Previous treatment with inhaled fluticasone furoate in a phase II or III study
* Current smokers or former smokers with significant tobacco exposure
* Children in Care

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (10):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Waco, Texas
- Mexico (3):
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Villahermosa, Tabasco
- Peru (3):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Borja, Lima region
  - GSK Investigational Site, San Miguel, Lima region
- Russia (6):
  - GSK Investigational Site, Klin
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- [Derived] O'Byrne PM, Woodcock A, Bleecker ER, Bateman ED, Lotvall J, Forth R, Medley H, Jacques L, Busse WW. Efficacy and safety of once-daily fluticasone furoate 50 mcg in adults with persistent asthma: a 12-week randomized trial. Respir Res. 2014 Aug 11;15(1):88. doi: 10.1186/s12931-014-0088-z. PMID 25108545
- [Derived] Svedsater H, Jacques L, Goldfrad C, Bleecker ER. Ease of use of the ELLIPTA dry powder inhaler: data from three randomised controlled trials in patients with asthma. NPJ Prim Care Respir Med. 2014 Jun 26;24:14019. doi: 10.1038/npjpcrm.2014.19. No abstract available. PMID 24966061
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 115283 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115283 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115283 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115283 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115283 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115283 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115283 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting eligibility criteria at the Screening visit entered a 2-week Run-in Period for Baseline safety evaluations and to obtain measures of asthma status. Participants were then randomized to a 12-week Treatment Period. A total of 449 participants were screened; 248 were randomized, and 242 received >=1 dose of study treatment.
Groups:
- Placebo: Participants receieved placebo via a Dry Powder Inhaler (DPI) once daily (OD) in the evening for 12 weeks. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 50 µg OD: Participants received fluticasone furoate (FF) 50 micrograms (µg) inhalation powder via a DPI OD in the evening for 12 weeks. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
Period: Overall Study
Arm/Group | Placebo | FF 50 µg OD
Started | 124 (These participants were randomized to trial medication.) | 124 (These participants were randomized to trial medication.)
Safety Population | 121 (These randomized participants received at least a single dose of trial medication.) | 121 (These randomized participants received at least a single dose of trial medication.)
Completed | 98 | 110
Not Completed | 26 | 14
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 16 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Did Not Receive Trial Medication | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 50 µg OD | Total
Number analyzed (Participants) | 121 | 121 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.5 (13.81) | 36.8 (15.98) | 35.2 (14.99)
Gender [Count of Participants; unit: Participants]
  Female | 75 | 70 | 145
  Male | 46 | 51 | 97
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 6 | 7 | 13
  American Indian or Alaska Native | 59 | 46 | 105
  Asian | 1 | 0 | 1
  White | 32 | 44 | 76
  African American/African Heritage & White | 2 | 0 | 2
  American Indian or Alaska Native & White | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Visit Evening (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at the End of the 12-week Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Evening clinic visit FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1 measurement taken at the Week 12 clinic visit. Pre-dose and pre-rescue albuterol/salbutamol trough FEV1 were measured electronically by spirometry in the evening at the Baseline through Week 12 clinic visits. The highest of 3 technically acceptable measurements was recorded. Baseline was the pre-dose value obtained at Visit 2. Change from Baseline was calculated as the Week 12 value minus the Baseline value. Analysis was performed using analysis of covariance (ANCOVA) with covariates of Baseline, region, sex, age, and treatment. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing, pre-dose, post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing value.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Population: all participants (par.) randomized to treatment who received >=1 dose of study medication, except for the par. of one investigator (excluded after good clinical practice [GCP] issues identified during a site audit). Only those par. with non-missing covariates and a post-Baseline FEV1 measurement were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 50 µg OD
Number analyzed (Participants) | 106 | 108
Liters | 0.038 (0.0333) | 0.157 (0.0330)
Statistical Analysis 1: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.012, ANCOVA; Median Difference (Final Values) = 0.120, 95% CI 2-sided [0.026 to 0.213]

2. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods Over the 12-week Treatment Period
Description: The number of inhalations of rescue bronchodilator, albuterol/salbutamol inhalation aerosol, used during the day and night was recorded by the participants in a daily electronic diary (eDiary). A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered to be rescue free. A 24-hour period was considered as missing if both day time and night time values were missing or if one of the day time or night time values were missing and the other value indicated no use of rescue medication. The Baseline value is the average of the values over the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | FF 50 µg OD
Number analyzed (Participants) | 110 | 111
Percentage of rescue-free 24-hr periods | 17.1 (2.78) | 28.7 (2.77)

3. Secondary Outcome: Change From Baseline in Daily Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the 12-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the average of the values of the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily trough PM PEF over the 12-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | Placebo | FF 50 µg OD
Number analyzed (Participants) | 110 | 111
Liters/minute (L/min) | 19.5 (3.72) | 22.8 (3.70)

4. Secondary Outcome: Change From Baseline in Daily Morning (AM) PEF Averaged Over the 12-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the average of the values of the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily AM PEF over the 12-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | FF 50 µg OD
Number analyzed (Participants) | 110 | 111
L/min | 22.9 (3.65) | 34.5 (3.64)

5. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods Over the 12-week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. A 24-hour period was considered as missing if both the day time and night time data were missing or if one was symptom-free but the other was missing. The Baseline value was the average of the values of the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 12-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | FF 50 µg OD
Number analyzed (Participants) | 110 | 111
Percentage of symptom-free 24-hr periods | 14.0 (2.49) | 22.6 (2.47)

6. Secondary Outcome: Number of Participants Who Withdrew Due to a Lack of Efficacy During the 12-week Treatment Period
Description: The reason for withdrawal was lack of efficacy if a participant was withdrawn due to: clinic FEV1 falling below the FEV1 stability limit; participant experiencing at least 4 days of AM or PM PEF falling below the PEF stability limit and/or at least 3 days of >=12 inhalations/day of albuterol/salbutamol usage during the 7 days immediately preceding any contact; or the occurrence of an asthma exacerbation, defined as the deterioration of asthma requiring the use of systemic (oral, parenteral, or depot) corticosteroids for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids. The FEV1 stability limit was calculated as the best pre-salbutamol/albuterol FEV1 at Visit 2 * 80%. The PEF stability limit was calculated as the mean AM PEF from the available 7 consecutive days preceding Visit 2 * 80%.
Time Frame: From the first dose of the study medication until Week 12/Early Withdrawal
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 50 µg OD
Number analyzed (Participants) | 111 | 111
Participants | 15 | 7

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs), defined as those events occurring while participants were on treatment, up to and including the day after the last dose (up to 12 weeks), are reported.
Description: Serious AEs (SAEs) and non-serious AEs were collected in the Safety Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | Placebo | FF 50 µg OD
Serious Adverse Events (participants affected / at risk) | 1/121 | 1/121
Other Adverse Events (participants affected / at risk) | 27/121 | 18/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | FF 50 µg OD (N=121)
Appendicitis perforated (Infections and infestations) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | FF 50 µg OD (N=121)
Nasopharyngitis (Infections and infestations) | 5 | 7
Pharyngitis (Infections and infestations) | 6 | 6
Influenza (Infections and infestations) | 4 | 1
Headache (Nervous system disorders) | 14 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.